CLINICAL TRIAL: NCT03339323
Title: The Effect of Exercise Training on Muscle Mass in Patients With Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Robert Wen-Wei Hsu, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CORPG6G0261-3
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Knee Osteoarthritis; Arthropathy of Knee Joint
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard rehabilitation procedure
- Exercise (Experimental): Aerobic exercise combined with resistance training; Concentric resistance training; Eccentric resistance training
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — TKA patients do the exercise intervention
  Arms: Exercise

SUMMARY:
Background:

Total knee arthroplasty (TKA) is one of the most common operations in orthopedics. After surgery, the decline of bone mineral density and muscle mass was proved, oral bisphosphonate is commonly used to prevent BMD loss in clinic treatment, however, the loss of muscle mass can only be maintained with exercise intervention. The goals of TKA rehabilitation should be based on control pain, improve ambulation, maximize the range of motion, develop muscle strength, and provide emotional support. We planned to find out a potential adjuvant effective option in muscle mass for the management of post-TKA. Literature suggested that exercise training has been found to have the considerable effect on TKA. However, no suitable exercise prescription was established on the scientific basis. The current study aimed to find out a potential treatment mode.

Study Rationale:

This project will be performed for consecutive three years, the patients with post-TKA patients are managed with the treadmill exercise training in the first year. In the second year, resistance exercise is prescribed. In the third year, eccentric exercise plus resistance training will be arranged in the exercise group. We will analyze the data of the three years and cross-comparative analysis. A prescription of exercise training, a period of 24 weeks each year, 3 times a week, for each 10 minutes warm-up, 40 minutes exercise training, and 10-minute cool down for exercise prescription

Study Objectives:

To investigate the effect of long-term exercise training, eccentric and resistance exercise on muscle mass in patients with total knee arthroplasty. To monitor the performance index included: physiological indices, muscle mass, ambulation and the quality of life index.

Study Design Duration of Treatment: Total of 6-month exercise intervention in each year. The number of Planned Patients: 35 subjects in each control and exercise group in one year, the total of 210 subjects in three years.

Investigational Product: Automated biochemistry analyzer, Biospace Inbody 7.20 Analysis of body composition instrumentation; Dual Energy X-ray Absorptiometer (DEXA), isokinetic muscle strength measurement, VICON to analysis ambulation, functional fitness, the questionnaire including SF-36, KOOS and VAS pain score.

Endpoints: Data collection in pre-surgery, 3 months, 6 months, 9 months and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of this study were the patients diagnosed with serious osteoarthritis (OA) and recommended to receive TKA surgery.

Exclusion Criteria:

* The exclusion criteria were the patients with Diabetes, Neuromusculoskeletal disorder, severe chronic disease, history of fracture of a lower limb, artificial limb, and unsuitable for exercise training

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline muscle mass | Baseline; three month ; six month and nine month after operation; twelve-month follow-up
  Muscle mass measurement is measured by dual-energy x-ray absorptiometry (DXA). DXA measures the muscle mass of the whole body and the measurement is assessed at pre-operation, three months, six months and nine months after the operation, and twelve-month follow-up.

SECONDARY OUTCOMES:
Change from baseline lower extremity muscle strength | Baseline; three month ; six month and nine month after operation; twelve-month follow-up
  Lower extremity muscle strength, including extension and flexion of the hip, knee and ankle were tested by the HUMAC NORM system (CSMi, Stoughton, MA) with the eccentric/concentric contraction mode at an angular velocity of 60 degrees/s.Isokinetic tests were performed five times for each participant, and each test was separated by a rest period of 3 min. The participants are assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up and received verbal encouragement during the exertion of peak torque.
Motion analysis | Baseline; three month ; six month and nine month after operation; twelve-month follow-up
  Gait analysis by VICON three-dimensional, 8-camera motion capture system.The outcome measurement is assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up.
Change from baseline SF-36 questionnaire assessment | Baseline; three month ; six month and nine month after operation; twelve-month follow-up
  SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower score the more disability. The higher the score the less disability. Eight sections including physical function, role limitation due to physical problems, bodily pain, general health, vitality, social functioning, role limitation due to emotional problems, and mental health. Additionally, the eight health domains can be used to provide a physical component summary and mental component summary score. The outcome measurement is assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up.
Change from baseline KOOS questionnaire assessment | Baseline; three month ; six month and nine month after operation; twelve-month follow-up
  KOOS contains 5 subscales with a total of 42 items: 1) pain, 2) other symptoms, 3) function in daily living (ADL), 4) function in sport and recreation and 5) knee-related quality of life. Each question receives a score from 0 to 4 and the scores are transformed to a 0-100 score (0, extreme symptoms, 100, no symptoms). The User's Guide, is available from www.koos.nu. The outcome measurement is assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up.
Physical fitness---6-minutes' walk test | Baseline; three month , six month and nine month after operation; twelve-month follow-up
  The 6-minutes' walk test measures the distance an individual is able to walk over a total of 6 minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in 6 minutes and is assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up.
Physical fitness---8 feet up and go | Baseline; three month , six month and nine month after operation; twelve-month follow-up
  The 8 feet up and go test indicates the level of the participant's motor agility and dynamic balance and is assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up.
Physical fitness---30-sec sit to stand | Baseline; three month , six month and nine month after operation; twelve-month follow-up
  30-sec sit to stand (times in 30sec) is assessed lower body strength, needed for numerous tasks such as climbing stairs, walking and getting out of a chair. Also reduces the chance of falling. Number of full stands that can be completed in 30 seconds with arms folded across chest and is assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Sports Medicine Center, Chang Gung Memorial Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided